CLINICAL TRIAL: NCT00577434
Title: The Pharmacokinetics and Pharmacodynamics of a Single Dose of Pentobarbital for Clinically Indicated Sedation for Neonates, Infants, and Children Recovering From Open Heart Surgery
Brief Title: Pharmacokinetics and Pharmacodynamics of Pentobarbital in Neonates, Infants, and Children Following Open Heart Surgery
Status: Terminated | Type: Observational
Why Stopped: Sluggish enrollment
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-4-4822; CTRC 2012
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2008-07

CONDITIONS: Cardiac Surgical Procedures
Keywords: Procedural sedation; Sedation for diagnostic imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This medication is used for procedural sedation and sedation for diagnostic imaging. The purpose of this study is to find out what happens to pentobarbital in the body after it is given to children who have had heart surgery.

DETAILED DESCRIPTION:
This clinical trial of pentobarbital admistered as a bolus dose for procedural or imaging seddation will determine the PK of the drug in neonates, infants,, and children who are postoperative from cardiac surgery. Pediatric patients hsopitalized in the CICU who would receive IV bolus doses of pentobarbital as standard of care are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Will receive intravenous pentobarbital for procedural/imaging sedation as standard of care
* Age(Neonates, Young Infants, Older Infants, and Children Up to 6 years old)
* Diagnosis either postop from cardiac surgery or requrie sedation with IV pentobarbital as standard of care
* Adequate liver function tests
* Informed consent

Exclusion Criteria:

* Pregnant or lactating females
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients enrolled in this study will be postoperative from cardiac surgery adn have require sedation for a procedure or diagnostic imaging.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athena Zuppa, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States